CLINICAL TRIAL: NCT00124280
Title: Open Label, Non-randomized, Phase 2 Study Investigating the Effect of RAD001 Monotherapy in Patients With Advanced NSCLC Previously Treated With Either Chemotherapy Only or With Chemotherapy and EGFR Inhibitor(s)
Brief Title: Study Investigating the Effect of Everolimus Monotherapy in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2235
Record Dates: First submitted 2005-07-26; First posted 2005-07-27 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Non-small-cell Lung Carcinoma
Keywords: Lung cancer; non-small cell; everolimus; Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Everolimus

ARMS (2):
- previously treated with chemotherapy only (Experimental): patients previously treated with chemotherapy only (at most 2 prior regimens one of which must have been platinum-based) and no EGFRI
  Interventions: Drug: RAD001
- previously treated with chemotherapy + small (Experimental): patients previously treated with chemotherapy (at most 2 prior regimens one of which must have been platinum-based) and with one small molecule EGFRI
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001
  Other Names: Everolimus

SUMMARY:
This study will evaluate the efficacy and safety of everolimus treatment of patients with advanced NSCLC. The rationale for investigating everolimus in advanced NSCLC previously treated with chemotherapy or chemotherapy plus EGFR inhibitors, like gefitinib or erlotinib, is based on following:

* The medical need for the better therapy for advanced NSCLC and limited efficacy of the currently available therapy in advanced NSCLC.
* Postulated association of relevant cell-signaling pathways targeted by everolimus with different aspects of oncogenesis, disease progression, and response/resistance to treatment.
* Effectiveness of everolimus and rapamycin in preclinical models of lung cancer
* Early reports of clinical responses to monotherapy with mTOR inhibitors in advanced NSCLC.

There is evidence that an enhanced PI3K/Akt/mTOR pathway, which is inhibited by everolimus, may be one of the key changes accounting for different aspects of oncogenesis, disease progression, and response/resistance to NSCLC cancer treatment. The use of the mTOR inhibitor everolimus in treatment of advanced NSCLC would be a novel therapeutic approach that proposes to logically manipulate the cell's regulatory pathways to enable control of tumor growth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced (unresectable or metastatic) NSCLC
* Tissue sample of the metastatic or primary tumor available for pathology evaluation and molecular marker analyses
* Patients who have received ≤ 2 chemotherapy regimens, one of which must have included cisplatinum or carboplatin, and who have documented evidence of tumor progression (Arm 1)
* Patients who have received ≤ 2 chemotherapy regimens, one of which must have included cisplatinum or carboplatin as well as a small molecule EGFR inhibitor (as a separate regimen) with documented tumor progression despite at least 4 weeks therapy with either gefitinib or erlotinib (Arm 2)

Exclusion Criteria:

* Concurrent therapy with agents used otherwise as anticancer therapy (for example, methotrexate for rheumatoid arthritis)
* Any investigational drug, other than EGFR inhibitor (Arm 2), within the preceding 4 weeks
* Chronic treatment with steroids or another immunosuppressive agent
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-07; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy based on the evaluation of objective tumor response rate (RR) | until progressive disease or unacceptable toxicity.

SECONDARY OUTCOMES:
To assess safety of RAD001 monotherapy | as long as patients are in the study
To assess additional clinical efficacy of RAD001 | as long as patients are in the study
To assess the steady state levels of RAD001 in blood | as long as patients are in the study
To investigate potential molecular markers predictive of clinical effect | as long as patients are in the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceutcals
Locations (2):
- United States (2):
  - Nevada Cancer Institute, Las Vegas, Nevada
  - MD Anderson Cancer Center, Department of Thoracic /Head and Neck Medical Oncology, Houston, Texas

REFERENCES:
- [Result] White DA, Schwartz LH, Dimitrijevic S, Scala LD, Hayes W, Gross SH. Characterization of pneumonitis in patients with advanced non-small cell lung cancer treated with everolimus (RAD001). J Thorac Oncol. 2009 Nov;4(11):1357-63. doi: 10.1097/JTO.0b013e3181ba20b1. PMID 19745764
- [Result] Soria JC, Shepherd FA, Douillard JY, Wolf J, Giaccone G, Crino L, Cappuzzo F, Sharma S, Gross SH, Dimitrijevic S, Di Scala L, Gardner H, Nogova L, Papadimitrakopoulou V. Efficacy of everolimus (RAD001) in patients with advanced NSCLC previously treated with chemotherapy alone or with chemotherapy and EGFR inhibitors. Ann Oncol. 2009 Oct;20(10):1674-81. doi: 10.1093/annonc/mdp060. Epub 2009 Jun 23. PMID 19549709